CLINICAL TRIAL: NCT04819386
Title: Prospective Pilot Study of the NEIVATECH Virtual Reality-based System to Improve Visual Function in Children with Amblyopia
Brief Title: NEIVATECH Virtual Reality-based System for Amblyopia
Acronym: NEIVATECH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Increase-Tech (Other)
Collaborators: University of Alicante (Other); University of Valladolid (Other); Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Principal Investigator, Juan Francisco Arenillas Lara, Principal Investigator, Increase-Tech
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASVE-NM-21-516
Record Dates: First submitted 2021-03-18; First posted 2021-03-29 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2023-09

CONDITIONS: Amblyopia
Keywords: Amblyopic children; Perceptual learning; Dichoptic training; Virtual reality; Gamification
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active group (Experimental): 18 half-hour in-office active vision therapy sessions with the NEIVATECH Virtual Reality-based system
  Interventions: Other: Active vision therapy sessions with the NEIVATECH Virtual Reality-based system

INTERVENTIONS:
Other: Active vision therapy sessions with the NEIVATECH Virtual Reality-based system — The active visual therapy sessions with the NEIVATECH Virtual Reality-based system will be 18 in total, will have an average duration of half an hour and will be distributed over a month as follows: 5 sessions in the first two weeks after enrollment (Monday to Friday) and 4 sessions in the next two weeks (Monday to Thursday).

SUMMARY:
The NEIVATECH system has been designed to provide binocular vision training to 7-15 year old amblyopic children by discriminating Gabor patches presented with different contrast to each eye as a perceptual learning task.

DETAILED DESCRIPTION:
Due to the global impact of amblyopia, there is a medical and social need, and at the same time, a clear market niche, for the design and development of new therapies that can improve recurrence rates and non-compliance with conventional treatments. In this sense, the aim of this single-arm, multicentre, prospective pilot study is to examine the safety, acceptability and clinical efficacy of a novel Virtual Reality-based system designed to provide binocular vision training to 7-15 year old amblyopic children complementing the concepts of perceptual learning and dichoptic training with a gamification approach.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 7 and 15 years.
* VA in the amblyopic eye < 0.1 logMAR units.
* Interocular difference in VA ≥ 1 logMAR line.
* Interocular difference in espherical equivalent ≥ 1 D.
* Interpupillary distance (IPD) between 60.7 and 73.5 mm.
* Use of best refractive correction for at least 2 months prior to inclusion.
* Lack of response or therapeutic adherence to conventional occlusion therapy.
* Willingness to attend all the active vision therapy sessions and/or visits of the study.
* No history of previous treatment for amblyopia other than optimal refractive correction for at least 2 months prior to inclusion.

Exclusion Criteria:

* Active eye disease.
* Previous ocular surgery.
* BCVA in the amblyopic eye of ≥ 0.70 logMAR.
* Presence of cognitive impairment or neurological or psychiatric disorders.
* Presence of irregular cornea due to astigmatism or ectatic corneal disease.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change in distance best-corrected visual acuity (BCVA) | Baseline - 1 month
  ETDRS, logMAR scale, maximum -0.3 (best) and minimum 1.20 (worse)

SECONDARY OUTCOMES:
Change in near BCVA | Baseline - 1 month
  ETDRS, logMAR scale, maximum -0.3 (best) and minimum 1.20 (worse)
Change in photopic contrast sensitivity function (CSF) | Baseline - 1 month
  CSV-1000 test for spatial frequencies of 3, 6, 12 and 18 cycles/degree

OTHER OUTCOMES:
Change in refraction under cycloplegia | Baseline - 1 month
  Magnitude of sphere and cylinder (diopters), orientation of axis of astigmatism (degrees)
Change in stereopsis | Baseline - 1 month
  Magnitude of stereoacuity (seconds of arc)
Change in binocular vision | Baseline - 1 month
  Worth's four dot test and Four prism dioptre reflex text
Change in fusional vergence | Baseline - 1 month
  Magnitude of base-out and base-in prisms needed to obtain diplopia while the patient is looking at a distance and near (40 cm) stimulus
Change in accommodative facility | Baseline - 1 month
  Number of changes performed achieving an optimum focus using a spherical flipper of +-2.00 D while the patient is looking at a near optotype (VA 0,63)
Change in near point of convergence | Baseline - 1 month
  Closest distance in cm in reference to the nasal root of the patient at which the subject is able to maintain single vision

CONTACTS AND LOCATIONS:
Overall Officials: Juan Francisco Arenillas Lara, PhD, Principal Investigator — University of Valladolid
Locations (2):
- Spain (2):
  - University Clinical Hospital of Valladolid, Valladolid, Valladolid
  - Vithas Medimar International Hospital, Alicante

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leal-Vega L, Coco-Martin M feminineB, Molina-Martin A, Cuadrado-Asensio R, Vallelado-Alvarez AI, Sanchez-Tocino H, Mayo-Iscar A, Hernandez-Rodriguez CJ, Arenillas Lara JF, Pinero DP. NEIVATECH pilot study: immersive virtual reality training in older amblyopic children with non-compliance or non-response to patching. Sci Rep. 2024 Nov 14;14(1):28062. doi: 10.1038/s41598-024-79565-y. PMID 39543340
- [Derived] Leal Vega L, Pinero DP, Hernandez Rodriguez CJ, Molina Martin A, Morales-Quezada L, Vallelado Alvarez AI, Arenillas Lara JF, Coco Martin MB. Study protocol for a randomized controlled trial of the NEIVATECH virtual reality system to improve visual function in children with anisometropic amblyopia. BMC Ophthalmol. 2022 Jun 7;22(1):253. doi: 10.1186/s12886-022-02466-z. PMID 35672688